CLINICAL TRIAL: NCT04031846
Title: A Phase 3, Multicenter, Randomized, Double-blind, Active-comparator-controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of V114 in Healthy Infants (PNEU-PED-EU-1)
Brief Title: Safety, Tolerability, and Immunogenicity of V114 in Healthy Infants (V114-025)
Acronym: PNEU-PED-EU-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V114-025; V114-025 (Other: Merck, Sharp & Dohme); 2018-003787-31 (EudraCT Number)
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — RIX4414 vaccine; 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- V114 (Experimental): Full-term infants received a 0.5 mL intramuscular injection of V114 at approximately 2, 4, and 11-15 months of age (Study Day 1, Month 2, and Month 9-13). Preterm infants received a 0.5 mL intramuscular injection of V114 at approximately 2, 3, 4, and 11-15 months of age (Study Day 1, Month 1, Month 2, and Month 9-13). All infants also received intramuscular injection of 0.5 mL Infanrix™ hexa at approximately 2, 3, 4, and 11-15 months of age and 1.5 mL oral dose of Rotarix™ at 2 and 4 months of age.
  Interventions: Drug: Rotarix™; Drug: Infanrix™ hexa; Drug: V114
- Prevenar 13™ (Active Comparator): Full-term infants received a 0.5 mL intramuscular injection of Prevenar 13™ at approximately 2, 4, and 11-15 months of age (Study Day 1, Month 2, and Month 9-13). Preterm infants received a 0.5 mL intramuscular injection of Prevenar 13™ at approximately 2, 3, 4, and 11-15 months of age (Study Day 1, Month 1, Month 2, and Month 9-13). All infants also received intramuscular injection of 0.5 mL Infanrix™ hexa at approximately 2, 3, 4, and 11-15 months of age and 1.5 mL oral dose of Rotarix™ at 2 and 4 months of age.
  Interventions: Drug: Rotarix™; Drug: Infanrix™ hexa; Drug: Prevenar 13™

INTERVENTIONS:
Drug: Rotarix™ — Single 1.5 mL oral dose at 2 and 4 months of age (Study Day 1 and Month 2)
Drug: Infanrix™ hexa — Single 0.5 mL intramuscular injection at 2, 3, 4, and 11-15 months of age (Study Day 1, Month 1, Month 2, and Month 9-13)
Drug: V114 — 15-valent pneumococcal conjugate vaccine (PCV) containing 13 serotypes present in Prevenar 13™ (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) and 2 unique serotypes (22F and 33F) in each 0.5 mL intramuscular administration,
  Other Names: VAXNEUVANCE™; Pneumococcal 15-Valent Conjugate Vaccine
  Arms: V114
Drug: Prevenar 13™ — 13-valent PCV containing 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) in each 0.5 mL intramuscular administration.
  Arms: Prevenar 13™

SUMMARY:
This study will evaluate the safety and tolerability and immunogenicity of V114 when administered to 2-month old infants. The primary hypotheses are: 1) V114 is non-inferior to Prevenar 13™ for the 13 shared serotypes between V114 and Prevenar 13™ based on response rates at 30 days post toddler dose (PTD); 2) V114 is superior to Prevenar 13™ for the 2 serotypes unique to V114 based on the response rates at 30 days PTD; 3) V114 is non-inferior to Prevenar 13™ for the 13 shared serotypes between V114 and Prevenar 13™ based on anti-pneumococcal polysaccharide (PnPs) serotype-specific Immunoglobin G (IgG) geometric mean concentrations (GMCs) at 30 days PTD; and 4) V114 is superior to Prevenar 13™ for the 2 serotypes unique to V114 based on anti-PnPs serotype-specific IgG GMCs at 30 days PTD.

ELIGIBILITY:
Inclusion Criteria

* Healthy
* Has a legally acceptable representative who understands the study procedures, alternate treatments available, and risks involved with the study and voluntarily agrees to participate by giving written informed consent

Exclusion Criteria

* History of invasive pneumococcal disease [(IPD); positive blood culture, positive cerebrospinal fluid culture, or other sterile site] or known history of other culture positive pneumococcal disease
* Has a known or suspected impairment of immunological function
* Has a history of congenital or acquired immunodeficiency
* Has, or his/her mother has, a documented human immunodeficiency virus (HIV) infection
* Has, or his/her mother has, a documented hepatitis B surface antigen - positive test
* Has known or history of functional or anatomic asplenia
* Has failure to thrive based on the clinical judgement of the Investigator
* Has a bleeding disorder contraindicating intramuscular vaccination
* Has a history of autoimmune disease (including but not limited to systemic lupus erythematosus, antiphospholipid syndrome, Behcet's disease, autoimmune thyroid disease, polymyositis and dermatomyositis, scleroderma, Type 1 diabetes mellitus, or other autoimmune disorders)
* Has a known neurologic or cognitive behavioral disorder, including encephalitis/myelitis, acute disseminating encephalomyelitis, pervasive development disorder, and related disorders
* Has received a dose of any pneumococcal vaccine prior to study entry
* Has received >1 dose of monovalent hepatitis B vaccine or hepatitis B-based combination vaccine prior to study entry
* Has received a dose of any acellular pertussis- or whole cell pertussis-based combination vaccines, Haemophilus influenzae type b conjugate vaccine, poliovirus vaccine, rotavirus vaccine, or any other combination thereof, prior to study entry
* Has received a blood transfusion or blood products, including immunoglobulins
* Has participated in another clinical study of an investigational product before the beginning or anytime during the duration of the current clinical study. Participants enrolled in observational studies may be included; these will be reviewed on a case-by-case basis for approval by the Sponsor
* Is or has an immediate family member (eg, parent/legal guardian or sibling) who is investigational site or Sponsor staff directly involved with this study

Ages: 42 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1184 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (60):
- Australia (3):
  - Queensland Children s Hospital ( Site 0004), South Brisbane, Queensland
  - Vaccine and Immunisation Research Group - VIRGo ( Site 0002), Melbourne, Victoria
  - Telethon Kids Institute ( Site 0003), Nedlands
- Belgium (6):
  - O.L.V. Ziekenhuis Aalst ( Site 0144), Aalst
  - AZ Sint Jan Brugge-Oostende ( Site 0147), Bruges
  - AZ Maria Middelares Gent ( Site 0142), Ghent
  - UZ Gent ( Site 0141), Ghent
  - AZ Henry Serruys ( Site 0148), Ostend
  - AZ Delta ( Site 0143), Roeselare
- Czechia (3):
  - MUDr. Daniel Drazan - Prakticky lekar pro deti a dorost ( Site 0151), Jindřichův Hradec
  - MU Dr. Jan Nemecek - Prakticky lekar pro deti a dorost ( Site 0152), Mělník
  - MUDr. Josef Zemanek ( Site 0153), Týnec nad Sázavou
- Estonia (6):
  - Vee Perearstikeskus ( Site 0163), Paide, Järvamaa
  - Merekivi Perearstid ( Site 0165), Tallinn
  - Merelahe Perearstikeskus OU ( Site 0164), Tallinn
  - Sinu Arst Tervisekeskus ( Site 0167), Tallinn
  - Rosenthali Perearstikeskus OU ( Site 0166), Tallinn
  - Kliiniliste Uuringute Keskus OU ( Site 0161), Tartu
- Germany (14):
  - NETSTAP - Sandner ( Site 0072), Aschaffenburg
  - Kinderarztpraxis ( Site 0061), Bramsche
  - Praxis Dr. Schmute ( Site 0078), Datteln
  - Praxis fur Kinder und Jugendmedizin Eivy Franke Beckmann ( Site 0064), Erfurt
  - Kinderarztpraxis Dr. Friedrich Kaiser & Dr. Marinesse ( Site 0065), Hamburg
  - Kinderarztpraxis Dr. Juenger ( Site 0073), Herxheim
  - Kinderpraxis Dr. med. Andreas Petri ( Site 0066), Hürth
  - Kinderarztpraxis ( Site 0068), Mönchengladbach
  - Kinder- und Jugendaerztliche Gemeinschaftspraxis ( Site 0077), Oberhausen
  - Praxiszentrum Triftplatz ( Site 0075), Schönau
  - Praxis Dr. Siegfried Simmet ( Site 0069), Schweigen
  - Kinderarztpraxis Dr. Rolf Ebert & Dr. Matthias Huebener ( Site 0062), Tauberbischofsheim
  - Kinderaerztliche Gemeinschaftspraxis Drs. Westerholt/Matyas ( Site 0074), Wolfsburg
  - Kinderarztpraxis ( Site 0063), Würselen
- Greece (5):
  - Pan and Aglaia Kyriakou Children s Hospital ( Site 0183), Athens
  - University of Athens - Aghia Sophia Childrens Hospital ( Site 0185), Athens
  - Attikon University General Hospital of Athens ( Site 0182), Athens
  - University General Hospital of Larissa ( Site 0184), Larissa
  - Hippokration General Hospital of Thessaloniki ( Site 0181), Thessaloniki
- Poland (9):
  - Centrum Medyczne Pratia Bydgoszcz ( Site 0086), Bydgoszcz
  - Prywatny Gabinet Lekarski Dr med Jerzy Brzostek ( Site 0084), Dębica
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II ( Site 0085), Krakow
  - Gravita Diagnostyka i Leczenie Nieplodnosci ( Site 0092), Lodz
  - SPZOZ Szpital Dzieciecy Poznan ( Site 0089), Poznan
  - NZ Lecznictwa Ambulatoryjnego - Michalkowice - Jarosz i Partnerzy ( Site 0087), Siemianowice Śląskie
  - Szpital im. sw. Jadwigi Slaskiej w Trzebnicy ( Site 0083), Trzebnica
  - Uniwersytecki Szpital Kliniczny ( Site 0093), Wroclaw
  - SPZOZ im. Dzieci Warszawy w Dziekanowie Lesnym ( Site 0091), Łomianki
- Russia (3):
  - Central Clinical Hospital of Russian Academy Science ( Site 0052), Moscow
  - Children s City Polyclinic No. 45 of the Nevsky District ( Site 0048), Saint Petersburg
  - MAI Childrens City Clinical Hospital 11 ( Site 0047), Yekaterinburg
- Spain (11):
  - Hospital Universitari Germans Trias i Pujol ( Site 0102), Badalona, Barcelona
  - Hospital de Antequera ( Site 0111), Antequera, Malaga
  - Centro de Salud Paiporta ( Site 0117), Paiporta, Valencia
  - C.S. Quart de Poblet ( Site 0115), Quart de Poblet, Valencia
  - Hospital General Universitario 12 de Octubre ( Site 0106), Madrid
  - Hospital Universitario La Paz ( Site 0107), Madrid
  - Hospital Sanitas La Moraleja ( Site 0103), Madrid
  - Hospital Clinico Universitario de Santiago ( Site 0109), Santiago de Compostela
  - Unidad de Estudios e Investigacion IHP ( Site 0101), Seville
  - C.S. Serreria II ( Site 0116), Valencia
  - Centro de Salud Eliana ( Site 0114), Valencia

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Martinon-Torres F, Wysocki J, Szenborn L, Carmona-Martinez A, Poder A, Dagan R, Richmond P, Gilbert C, Trudel MC, Flores S, Lupinacci R, McFetridge R, Wiedmann RT, Chen Q, Gerrits H, Banniettis N, Musey L, Bickham K, Kaminski J; V114-025 PNEU-PED-EU-1 study group. A Phase III, multicenter, randomized, double-blind, active comparator-controlled study to evaluate the safety, tolerability, and immunogenicity of V114 compared with PCV13 in healthy infants (PNEU-PED-EU-1). Vaccine. 2023 May 16;41(21):3387-3398. doi: 10.1016/j.vaccine.2023.04.036. Epub 2023 Apr 25. PMID 37105892

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Healthy males and females aged 42 to 90 days (inclusive) were enrolled. One participant randomized to the V114 group, who was cross-treated with both pneumococcal conjugate vaccines (PCVs), V114 and Prevenar 13™, was excluded from the all participants as treated (APaT) i.e. the safety endpoints population; but was included in the AE module as a separate treatment group.
Groups:
- V114: Full-term infants received a 0.5 mL intramuscular injection of V114 at approximately 2, 4, and 11-15 months of age (Study Day 1, Month 2, and Month 9-13). Preterm infants received a 0.5 mL intramuscular injection of V114 at approximately 2, 3, 4,and 11-15 months of age (Study Day 1, Month 1, Month 2, and Month 9-13). All infants also received licensed background intramuscular injections of 0.5 mL Infanrix™ hexa at approximately 2, 3, 4, and 11-15 months of age (Study Day 1, Months 1, 2, and Month 9-13); and also 1.5 mL oral dose of Rotarix™ at 2 and 4 months of age (Study Day 1 and Month 2).
- Prevenar 13™: Full-term infants received a 0.5 mL intramuscular injection of Prevenar 13™ at approximately 2, 4, and 11-15 months of age (Study Day 1, Month 2, and Month 9-13). Preterm infants received a 0.5 mL intramuscular injection of Prevenar 13™ at approximately 2, 3, 4, and 11-15 months of age (Study Day 1, Month 1, Month 2, and Month 9-13). All infants also received licensed background intramuscular injections of 0.5 mL Infanrix™ hexa at approximately 2, 3, 4, and 11-15 months of age (Study Day 1, Months 1, 2, and Month 9-13); and also 1.5 mL oral dose of Rotarix™ at 2 and 4 months of age (Study Day 1 and Month 2).
Period: Overall Study
Arm/Group | V114 | Prevenar 13™
Started | 591 | 593
Vaccinated | 588 (One participant was vaccinated with Prevenar 13™) | 591
All Participants As Treated | 587 (Excluded one vaccinated with Prevenar 13™) | 591
PCV Dose at Age 2 Months | 588 | 591
PCV Dose at Age 3 Months | 32 | 35
PCV Dose at Age 4 Months | 582 | 584
PCV Dose at Age 11-15 Months | 571 | 574
Completed | 569 | 570
Not Completed | 22 | 23
Not completed — Lost to Follow-up | 4 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal By Parent/Guardian | 17 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V114 | Prevenar 13™ | Total
Number analyzed (Participants) | 591 | 593 | 1184
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.4 (1.5) | 8.5 (1.5) | 8.5 (1.5)
Age, Customized [Number; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 591 | 593 | 1184
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0
  Adults (18-64 years) | 0 | 0 | 0
  From 65-84 years | 0 | 0 | 0
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 283 | 286 | 569
  Male | 308 | 307 | 615
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 66 | 65 | 131
  Not Hispanic or Latino | 525 | 526 | 1051
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 5 | 9
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 574 | 573 | 1147
  More than one race | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Report at Least 1 Solicited Injection-site Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of a study intervention. Injection-site AEs solicited on the Vaccine Report Card (VRC) consisted of erythema (redness), induration (hard lump), pain (tenderness) and swelling.
Time Frame: Up to 14 days post any vaccination (up to approximately study month 13)
Population: Participants who received at least 1 dose of study vaccination based on the group to which they were randomized, and corresponding to the study vaccination they actually received. One participant randomized to V114, who inadvertently received both V114 and Prevenar 13™, was excluded from this analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 587 | 591
Percentage of Participants
  Injection site erythema | 45.3 | 44.7
  Injection site induration | 41.9 | 39.1
  Injection site pain | 40.5 | 29.3
  Injection site swelling | 33.6 | 29.4
Statistical Analysis 1: Comparison: V114 vs Prevenar 13™; Difference in % : Injection site erythema; Test type: Other — Difference in % and 95 % confidence interval (CI) are calculated based on the Miettinen & Nurminen method; p = 0.824, Miettinen & Nurminen; Percentage Difference = 0.6, 95% CI 2-sided [-5.0 to 6.3] — V114 minus Prevenar 13™
Statistical Analysis 2: Comparison: V114 vs Prevenar 13™; Difference in %: Injection site induration; Test type: Other — Difference in % and 95 % CI are calculated based on the Miettinen & Nurminen method; p = 0.324, Miettinen & Nurminen; Percentage Difference = 2.8, 95% CI 2-sided [-2.8 to 8.4] — V114 minus Prevenar 13™
Statistical Analysis 3: Comparison: V114 vs Prevenar 13™; Difference in %: Injection site pain; Test type: Other — Difference in % and 95 % CI are calculated based on the Miettinen & Nurminen method; p < 0.001, Miettinen & Nurminen; Percentage Difference = 11.3, 95% CI 2-sided [5.8 to 16.6] — V114 minus Prevenar 13™
Statistical Analysis 4: Comparison: V114 vs Prevenar 13™; Difference in %: Injection site swelling; Test type: Other — Difference in % and 95 % CI are calculated based on the Miettinen & Nurminen method; p = 0.128, Miettinen & Nurminen; Percentage Difference = 4.1, 95% CI 2-sided [-1.2 to 9.4] — V114 minus Prevenar 13™

2. Primary Outcome: Percentage of Participants That Report at Least 1 Solicited Systemic AE
Description: An AE is any untoward medical occurrence in a participant temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of a study intervention. Systemic AEs solicited on the VRC consisted of decreased appetite (loss of appetite), irritability, somnolence (drowsiness) and urticaria (hive/welts).
Time Frame: Up to 14 days post any vaccination (up to approximately study month 13)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 587 | 591
Percentage of Participants
  Decreased appetite | 33.9 | 33.5
  Irritability | 71.7 | 66.3
  Somnolence | 46.2 | 41.8
  Urticaria | 3.7 | 3.9
Statistical Analysis 1: Comparison: V114 vs Prevenar 13™; Difference in %: Decreased appetite; Test type: Other — Difference in % and 95 % CI are calculated based on the Miettinen & Nurminen method; p = 0.885, Miettinen & Nurminen; Percentage Difference = 0.4, 95% CI 2-sided [-5.0 to 5.8] — V114 minus Prevenar 13™
Statistical Analysis 2: Comparison: V114 vs Prevenar 13™; Difference in %: Irritability; Test type: Other — Difference in % and 95 % CI are calculated based on the Miettinen & Nurminen method; p = 0.045, Miettinen & Nurminen; Percentage Difference = 5.4, 95% CI 2-sided [0.1 to 10.7] — V114 minus Prevenar 13™
Statistical Analysis 3: Comparison: V114 vs Prevenar 13™; Difference in %: Somnolence; Test type: Other — Difference in % and 95 % CI are calculated based on the Miettinen & Nurminen method; p = 0.131, Miettinen & Nurminen; Percentage Difference = 4.4, 95% CI 2-sided [-1.3 to 10.0] — V114 minus Prevenar 13™
Statistical Analysis 4: Comparison: V114 vs Prevenar 13™; Difference in %: Urticaria; Test type: Other — Difference in % and 95 % CI are calculated based on the Miettinen & Nurminen method; p = 0.898, Miettinen & Nurminen; Percentage Difference = -0.1, 95% CI 2-sided [-2.4 to 2.1] — V114 minus Prevenar 13™

3. Primary Outcome: Percentage of Participants That Report at Least 1 Vaccine-related Serious Adverse Event (SAE)
Description: A serious adverse event (SAE) is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, is a cancer, is an overdose, or is another important medical event. The relatedness of a vaccine to a SAE is determined by an investigator who is a qualified physician.
Time Frame: Up to 6 months post last vaccination (up to approximately study month 20)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 587 | 591
Percentage of Participants | 0.0 | 0.2
Statistical Analysis 1: Comparison: V114 vs Prevenar 13™; Difference in %; Test type: Other — Difference in % and 95 % CI are calculated based on the Miettinen & Nurminen method; Percentage Difference = -0.2, 95% CI 2-sided [-1.0 to 0.5] — V114 minus Prevenar 13™

4. Primary Outcome: Anti-pneumococcal Polysaccharide (PnPs) Serotype-specific Immunoglobin G (IgG) Geometric Mean Concentrations (GMC) for Each Serotype at 30 Days Post Toddler Dose (PTD)
Description: Sera from participants was used to measure vaccine-induced anti-PnPs serotype-specific IgG for each serotype using pneumococcal electrochemiluminescence (PnECL). The Geometric Mean Concentration (GMC) for each of the 13 serotypes shared by both V114 and Prevenar 13™ (Serotypes 1 to 23F); and the 2 serotypes unique to V114 (Serotypes 22F and 33F) was assessed. Per protocol, within-group CIs were not calculated.
Time Frame: 30 days PTD (Up to approximately study month 14)
Population: All randomized participants without deviations from the protocol that may substantially affect the results. Deviations include, but are not limited to, failure to receive vaccination; receipt of prohibited medication or vaccine; failure to receive vaccination at the required time point; failure to receive the required vaccination dose; and collection of blood sample at a time point outside of the prespecified time window.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 588 | 591
μg/mL
  Serotype 1: number analyzed (Participants) | 539 | 537
  Serotype 1 | 1.29 [NA to NA] — NA means that per protocol, no within-group measures of dispersion (MOD) were planned or calculated. | 2.08 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 3: number analyzed (Participants) | 539 | 537
  Serotype 3 | 0.84 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.66 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 4: number analyzed (Participants) | 539 | 535
  Serotype 4 | 1.29 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.73 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 5: number analyzed (Participants) | 539 | 535
  Serotype 5 | 1.97 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3.06 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 6A: number analyzed (Participants) | 539 | 535
  Serotype 6A | 3.10 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4.57 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 6B: number analyzed (Participants) | 539 | 535
  Serotype 6B | 4.17 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4.37 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 7F: number analyzed (Participants) | 539 | 536
  Serotype 7F | 3.09 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3.93 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 9V: number analyzed (Participants) | 539 | 537
  Serotype 9V | 2.14 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2.99 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 14: number analyzed (Participants) | 539 | 537
  Serotype 14 | 5.26 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 7.04 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 18C: number analyzed (Participants) | 539 | 536
  Serotype 18C | 1.94 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2.22 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 19A: number analyzed (Participants) | 539 | 535
  Serotype 19A | 4.68 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5.65 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 19F: number analyzed (Participants) | 539 | 537
  Serotype 19F | 4.09 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4.63 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 23F: number analyzed (Participants) | 538 | 535
  Serotype 23F | 1.52 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.75 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 22F: number analyzed (Participants) | 539 | 535
  Serotype 22F | 5.98 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.08 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 33F: number analyzed (Participants) | 539 | 530
  Serotype 33F | 3.41 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.07 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
Statistical Analysis 1: Comparison: V114 vs Prevenar 13™; Serotype 1 GMC Ratio: CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — Non-inferiority of V114 to Prevenar 13™ is based on the lower bound of the 2-sided 95% CI for the GMC ratio (V114/Prevenar 13™) being >0.5 (1-sided p-value <0.025); p < 0.001, t-distribution — 1-sided p-value; GMC Ratio = 0.62, 95% CI 2-sided [0.57 to 0.68] — V114/Prevenar 13™
Statistical Analysis 2: Comparison: V114 vs Prevenar 13™; Serotype 3 GMC Ratio: CI and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, t-distribution — 1-sided p-value; GMC Ratio = 1.28, 95% CI 2-sided [1.17 to 1.39] — V114/Prevenar 13™
Statistical Analysis 3: Comparison: V114 vs Prevenar 13™; Serotype 4 GMC Ratio: CI and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, t-distribution — 1-sided p-value; GMC Ratio = 0.75, 95% CI 2-sided [0.68 to 0.82] — V114/Prevenar 13™
Statistical Analysis 4: Comparison: V114 vs Prevenar 13™; Serotype 5 GMC Ratio: CI and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, t-distribution — 1-sided p-value; GMC Ratio = 0.64, 95% CI 2-sided [0.59 to 0.70] — V114/Prevenar 13™
Statistical Analysis 5: Comparison: V114 vs Prevenar 13™; Serotype 6A GMC Ratio: CI and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, t-distribution — 1-sided p-value; GMC Ratio = 0.68, 95% CI 2-sided [0.61 to 0.76] — V114/Prevenar 13™
Statistical Analysis 6: Comparison: V114 vs Prevenar 13™; Serotype 6B GMC Ratio: CI and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, t-distribution — 1-sided p-value; GMC Ratio = 0.95, 95% CI 2-sided [0.85 to 1.07] — V114/Prevenar 13™
Statistical Analysis 7: Comparison: V114 vs Prevenar 13™; Serotype 7F GMC Ratio: CI and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, t-distribution — 1-sided p-value; GMC Ratio = 0.79, 95% CI 2-sided [0.72 to 0.85] — V114/Prevenar 13™
Statistical Analysis 8: Comparison: V114 vs Prevenar 13™; Serotype 9V GMC Ratio: CI and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, t-distribution — 1-sided p-value; GMC Ratio = 0.72, 95% CI 2-sided [0.66 to 0.78] — V114/Prevenar 13™
Statistical Analysis 9: Comparison: V114 vs Prevenar 13™; Serotype 14 GMC Ratio: CI and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, t-distribution — 1-sided p-value; GMC Ratio = 0.75, 95% CI 2-sided [0.67 to 0.83] — V114/Prevenar 13™
Statistical Analysis 10: Comparison: V114 vs Prevenar 13™; Serotype 18C GMC Ratio: CI and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, t-distribution — 1-sided p-value; GMC Ratio = 0.88, 95% CI 2-sided [0.80 to 0.95] — V114/Prevenar 13™
Statistical Analysis 11: Comparison: V114 vs Prevenar 13™; Serotype 19A GMC Ratio: CI and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, t-distribution — 1-sided p-value; GMC Ratio = 0.83, 95% CI 2-sided [0.75 to 0.91] — V114/Prevenar 13™
Statistical Analysis 12: Comparison: V114 vs Prevenar 13™; Serotype 19F GMC Ratio: CI and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, t-distribution — 1-sided p-value; GMC Ratio = 0.88, 95% CI 2-sided [0.80 to 0.97] — V114/Prevenar 13™
Statistical Analysis 13: Comparison: V114 vs Prevenar 13™; Serotype 23F GMC Ratio: CI and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, t-distribution — 1-sided p-value; GMC Ratio = 0.87, 95% CI 2-sided [0.79 to 0.97] — V114/Prevenar 13™
Statistical Analysis 14: Comparison: V114 vs Prevenar 13™; Serotype 22F GMC Ratio: CI and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Superiority — Superiority of V114 to Prevenar 13™ is based on the lower bound of the 2-sided 95% CI for the GMC ratio (V114/Prevenar 13™) being >2.0 (1-sided p-value <0.025); p < 0.001, t-distribution — 1-sided p-value; GMC Ratio = 71.79, 95% CI 2-sided [65.16 to 79.10] — V114/Prevenar 13™
Statistical Analysis 15: Comparison: V114 vs Prevenar 13™; Serotype 33F GMC Ratio: CI and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Superiority — [test comment as in outcome 4, analysis 14]; p < 0.001, t-distribution — 1-sided p-value; GMC Ratio = 46.58, 95% CI 2-sided [42.19 to 51.42] — V114/Prevenar 13™

5. Primary Outcome: Percentage of Participants Who Meet Serotype-specific IgG Threshold Value of ≥0.35 μg/mL for Each Serotype at 30 Days PTD
Description: Sera from participants was used to measure vaccine-induced anti-PnPs serotype-specific IgG for the 15 serotypes using pneumococcal electrochemiluminescence (PnECL). The percentage of participants that achieve the threshold value of ≥0.35 μg/mL for each of the 13 serotypes shared by both V114 and Prevenar 13™ (Serotypes 1 to 23F); and the 2 serotypes unique to V114 (Serotypes 22F and 33F) was assessed.
Time Frame: 30 days PTD (Up to approximately study month 14)
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 588 | 591
Percentage of Participants
  Serotype 1: number analyzed (Participants) | 539 | 537
  Serotype 1 | 96.7 | 99.4
  Serotype 3: number analyzed (Participants) | 539 | 537
  Serotype 3 | 92.0 | 83.8
  Serotype 4: number analyzed (Participants) | 539 | 535
  Serotype 4 | 95.7 | 97.9
  Serotype 5: number analyzed (Participants) | 539 | 535
  Serotype 5 | 99.1 | 100.0
  Serotype 6A: number analyzed (Participants) | 539 | 535
  Serotype 6A | 98.5 | 98.9
  Serotype 6B: number analyzed (Participants) | 539 | 535
  Serotype 6B | 97.4 | 99.1
  Serotype 7F: number analyzed (Participants) | 539 | 536
  Serotype 7F | 99.8 | 99.8
  Serotype 9V: number analyzed (Participants) | 539 | 537
  Serotype 9V | 98.9 | 100.0
  Serotype 14: number analyzed (Participants) | 539 | 537
  Serotype 14 | 99.8 | 100.0
  Serotype 18C: number analyzed (Participants) | 539 | 536
  Serotype 18C | 98.9 | 99.3
  Serotype 19A: number analyzed (Participants) | 539 | 535
  Serotype 19A | 99.1 | 100.0
  Serotype 19F: number analyzed (Participants) | 539 | 537
  Serotype 19F | 99.6 | 100.0
  Serotype 23F: number analyzed (Participants) | 538 | 535
  Serotype 23F | 96.8 | 97.4
  Serotype 22F: number analyzed (Participants) | 539 | 535
  Serotype 22F | 99.6 | 5.8
  Serotype 33F: number analyzed (Participants) | 539 | 530
  Serotype 33F | 99.1 | 4.2
Statistical Analysis 1: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 1; Test type: Non-Inferiority — Non-inferiority of V114 to Prevenar 13™ is based on the lower bound of the 95% CI for the difference in percentages (V114 - Prevenar 13™) being >-10 percentage points (1-sided p-value <0.025); p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = -2.8, 95% CI 2-sided [-4.7 to -1.3] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 2: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 3; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = 8.2, 95% CI 2-sided [4.4 to 12.2] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 3: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 4; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = -2.2, 95% CI 2-sided [-4.5 to -0.1] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 4: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 5; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = -0.9, 95% CI 2-sided [-2.2 to -0.2] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 5: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 6A; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = -0.4, 95% CI 2-sided [-1.9 to 1.1] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 6: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 6B; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = -1.7, 95% CI 2-sided [-3.5 to -0.1] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 7: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 7F; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = 0.0, 95% CI 2-sided [-0.9 to 0.9] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 8: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 9V; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = -1.1, 95% CI 2-sided [-2.4 to -0.4] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 9: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 14; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = -0.2, 95% CI 2-sided [-1.0 to 0.5] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 10: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 18C; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = -0.4, 95% CI 2-sided [-1.8 to 0.9] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 11: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 19A; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = -0.9, 95% CI 2-sided [-2.2 to -0.2] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 12: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 19F; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = -0.4, 95% CI 2-sided [-1.3 to 0.3] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 13: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 23F; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = -0.5, 95% CI 2-sided [-2.7 to 1.5] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 14: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 22F; Test type: Superiority — Superiority of V114 to Prevenar 13™ is based on the lower bound of the 95% CI for the difference in percentages (V114 - Prevenar 13™) being >10 percentage points (1-sided p-value <0.025); p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = 93.8, 95% CI 2-sided [91.5 to 95.6] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 15: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 33F; Test type: Superiority — [test comment as in outcome 5, analysis 14]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = 94.9, 95% CI 2-sided [92.7 to 96.5] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method

6. Secondary Outcome: Percentage of Participants Who Meet Antigen-Specific Threshold Value for Each Antigen in Infanrix™ Hexa at 30 Days PTD
Description: Sera from participants was used to measure vaccine-induced responses to 10 pre-specified Infanrix™ hexa antigens with the following threshold (% ≥) values: Diphtheria toxoid-0.1 international unit (IU)/mL;Tetanus toxoid-0.1 IU/mL; Pertussis pertussis toxin (PT)-5 endotoxin unit (EU)/mL; Pertussis filamentous hemagglutinin (FHA)-5 EU/mL; Pertussis pertactin (PRN)-5 EU/mL; Haemophilus influenzae type b (Hib) polyribosylribitol phosphate (PRP)-0.15 μg/mL; hepatitis B surface antigen (HBsAg)-10 mIU/mL; Poliovirus 1,2 and 3-1:8 neutralizing antibodies (NAb) dilution.
Time Frame: 30 days PTD (Up to approximately study month 14)
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 588 | 591
Percentage of Participants
  Diphtheria toxoid: number analyzed (Participants) | 537 | 533
  Diphtheria toxoid | 99.3 | 99.8
  Tetanus toxoid: number analyzed (Participants) | 537 | 533
  Tetanus toxoid | 99.6 | 100.0
  Pertussis PT: number analyzed (Participants) | 537 | 533
  Pertussis PT | 99.4 | 99.6
  Pertussis FHA: number analyzed (Participants) | 537 | 533
  Pertussis FHA | 99.8 | 100.0
  Pertussis PRN: number analyzed (Participants) | 537 | 533
  Pertussis PRN | 99.6 | 100.0
  Hib PRP: number analyzed (Participants) | 524 | 523
  Hib PRP | 98.5 | 98.1
  HBsAg: number analyzed (Participants) | 522 | 521
  HBsAg | 99.2 | 100.0
  Poliovirus 1: number analyzed (Participants) | 526 | 521
  Poliovirus 1 | 100.0 | 100.0
  Poliovirus 2: number analyzed (Participants) | 525 | 525
  Poliovirus 2 | 100.0 | 100.0
  Poliovirus 3: number analyzed (Participants) | 531 | 523
  Poliovirus 3 | 100.0 | 99.8
Statistical Analysis 1: Comparison: V114 vs Prevenar 13™; Percentage Difference: Diphtheria toxoid; Test type: Non-Inferiority — Non-inferiority of Infanrix™ hexa administered concomitantly with V114 to Infanrix™ hexa administered concomitantly with Prevenar 13™ is based on the lower bound of the 2-sided 95% CI for the difference in percentages (V114 - Prevenar 13™) being greater than the -10% specified non-inferiority margin (1-sided p-value <0.025); p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = -0.6, 95% CI 2-sided [-1.7 to 0.4] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 2: Comparison: V114 vs Prevenar 13™; Percentage Difference: Tetanus toxoid; Test type: Non-Inferiority — Non-inferiority of Infanrix™ hexa administered concomitantly with V114 to Infanrix™ hexa administered concomitantly with Prevenar 13™ is based on the lower bound of the 2-sided 95% CI for the difference in percentages (V114 - Prevenar 13™) being greater than the -5% specified non-inferiority margin (1-sided p-value <0.025); p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = -0.4, 95% CI 2-sided [-1.3 to 0.3] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 3: Comparison: V114 vs Prevenar 13™; Percentage Difference: Pertussis PT; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = -0.2, 95% CI 2-sided [-1.3 to 0.9] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 4: Comparison: V114 vs Prevenar 13™; Percentage Difference: Pertussis FHA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = -0.2, 95% CI 2-sided [-1.0 to 0.5] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 5: Comparison: V114 vs Prevenar 13™; Percentage Difference: Pertussis PRN; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = -0.4, 95% CI 2-sided [-1.3 to 0.3] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 6: Comparison: V114 vs Prevenar 13™; Percentage Difference: Hib PRP; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = 0.4, 95% CI 2-sided [-1.3 to 2.1] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 7: Comparison: V114 vs Prevenar 13™; Percentage Difference: HBsAg; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = -0.8, 95% CI 2-sided [-2.0 to -0.0] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 8: Comparison: V114 vs Prevenar 13™; Percentage Difference: Poliovirus 1; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = 0.0, 95% CI 2-sided [-0.7 to 0.7] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 9: Comparison: V114 vs Prevenar 13™; Percentage Difference: Poliovirus 2; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = 0.0, 95% CI 2-sided [-0.7 to 0.7] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method
Statistical Analysis 10: Comparison: V114 vs Prevenar 13™; Percentage Difference: Poliovirus 3; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; p < 0.001, Miettinen & Nurminen — 1-sided p-value; Percentage Difference = 0.2, 95% CI 2-sided [-0.5 to 1.1] — V114 minus Prevenar 13™; 95% CI is based on the Miettinen & Nurminen method

7. Secondary Outcome: Anti-rotavirus Immunoglobulin A (IgA) Geometric Mean Titers (GMTs) at 30 Days Post Primary Series (PPS) of Rotarix™
Description: Sera from participants was used to measure vaccine-induced antibodies in response to vaccination with Rotarix™ by assessing the GMT for IgA. Per protocol, within-group CIs were not calculated.
Time Frame: 30 days PPS (Up to approximately study month 3)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 520 | 503
Titer | 45.39 [NA to NA] — NA means that per protocol, no within-group measures of dispersion (MOD) were planned or calculated. | 47.07 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
Statistical Analysis 1: Comparison: V114 vs Prevenar 13™; GMT Ratio: CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — Non-inferiority of Rotarix™ administered concomitantly with V114 to Rotarix™ administered concomitantly with Prevenar 13™ is based on the lower bound of the 2-sided 95% CI for the GMT ratio (V114/Prevenar 13™) being >0.5 (1-sided p-value <0.025); p < 0.001, t-distribution — 1-sided p-value; GMT Ratio = 0.96, 95% CI 2-sided [0.80 to 1.16] — V114/Prevenar 13™

8. Secondary Outcome: Anti-PnPs Serotype-specific IgG GMCs for Each Serotype at 30 Days PPS
Description: Sera from participants was used to measure vaccine-induced anti-PnPs serotype-specific IgG for each serotype using PnECL. The GMC for each of the 13 serotypes shared by both V114 and Prevenar 13™ (Serotypes 1 to 23F); and the 2 serotypes unique to V114 (Serotypes 22F and 33F) was assessed. Per protocol, within-group CIs were not calculated.
Time Frame: 30 days PPS (Up to approximately study month 3)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 588 | 591
μg/mL
  Serotype 1: number analyzed (Participants) | 522 | 500
  Serotype 1 | 1.30 [NA to NA] — NA means that per protocol, no within-group measures of dispersion (MOD) were planned or calculated. | 1.62 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 3: number analyzed (Participants) | 522 | 500
  Serotype 3 | 0.88 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.48 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 4: number analyzed (Participants) | 522 | 500
  Serotype 4 | 1.41 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.30 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 5: number analyzed (Participants) | 522 | 500
  Serotype 5 | 0.89 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.06 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 6A: number analyzed (Participants) | 522 | 500
  Serotype 6A | 0.64 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.42 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 6B: number analyzed (Participants) | 522 | 499
  Serotype 6B | 0.43 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.36 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 7F: number analyzed (Participants) | 522 | 500
  Serotype 7F | 2.04 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2.46 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 9V: number analyzed (Participants) | 522 | 500
  Serotype 9V | 1.23 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.43 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 14: number analyzed (Participants) | 522 | 500
  Serotype 14 | 3.87 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5.14 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 18C: number analyzed (Participants) | 522 | 500
  Serotype 18C | 1.17 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.37 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 19A: number analyzed (Participants) | 522 | 500
  Serotype 19A | 1.71 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2.20 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 19F: number analyzed (Participants) | 522 | 500
  Serotype 19F | 2.63 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3.40 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 23F: number analyzed (Participants) | 522 | 499
  Serotype 23F | 0.76 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.62 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 22F: number analyzed (Participants) | 522 | 500
  Serotype 22F | 2.76 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.05 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 33F: number analyzed (Participants) | 522 | 500
  Serotype 33F | 0.31 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.05 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
Statistical Analysis 1: Comparison: V114 vs Prevenar 13™; GMC Ratio Serotype 1: CI are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Other; GMC Ratio = 0.80, 95% CI 2-sided [0.73 to 0.88] — V114 / Prevenar 13™
Statistical Analysis 2: Comparison: V114 vs Prevenar 13™; GMC Ratio Serotype 3: CI are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Other; GMC Ratio = 1.85, 95% CI 2-sided [1.70 to 2.02] — V114 / Prevenar 13™
Statistical Analysis 3: Comparison: V114 vs Prevenar 13™; GMC Ratio Serotype 4: CI are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Other; GMC Ratio = 1.08, 95% CI 2-sided [0.98 to 1.19] — V114 / Prevenar 13™
Statistical Analysis 4: Comparison: V114 vs Prevenar 13™; GMC Ratio Serotype 5: CI are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Other; GMC Ratio = 0.84, 95% CI 2-sided [0.74 to 0.94] — V114 / Prevenar 13™
Statistical Analysis 5: Comparison: V114 vs Prevenar 13™; GMC Ratio Serotype 6A: CI are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Other; GMC Ratio = 0.45, 95% CI 2-sided [0.40 to 0.52] — V114 / Prevenar 13™
Statistical Analysis 6: Comparison: V114 vs Prevenar 13™; GMC Ratio Serotype 6B: CI are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Other; GMC Ratio = 1.18, 95% CI 2-sided [1.00 to 1.41] — V114 / Prevenar 13™
Statistical Analysis 7: Comparison: V114 vs Prevenar 13™; GMC Ratio Serotype 7F: CI are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Other; GMC Ratio = 0.83, 95% CI 2-sided [0.76 to 0.91] — V114 / Prevenar 13™
Statistical Analysis 8: Comparison: V114 vs Prevenar 13™; GMC Ratio Serotype 9V: CI are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Other; GMC Ratio = 0.86, 95% CI 2-sided [0.77 to 0.96] — V114 / Prevenar 13™
Statistical Analysis 9: Comparison: V114 vs Prevenar 13™; GMC Ratio Serotype 14: CI are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Other; GMC Ratio = 0.75, 95% CI 2-sided [0.66 to 0.86] — V114 / Prevenar 13™
Statistical Analysis 10: Comparison: V114 vs Prevenar 13™; GMC Ratio Serotype 18C: CI are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Other; GMC Ratio = 0.85, 95% CI 2-sided [0.77 to 0.95] — V114 / Prevenar 13™
Statistical Analysis 11: Comparison: V114 vs Prevenar 13™; GMC Ratio Serotype 19A: CI are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Other; GMC Ratio = 0.78, 95% CI 2-sided [0.70 to 0.87] — V114 / Prevenar 13™
Statistical Analysis 12: Comparison: V114 vs Prevenar 13™; GMC Ratio Serotype 19F: CI are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Other; GMC Ratio = 0.77, 95% CI 2-sided [0.70 to 0.85] — V114 / Prevenar 13™
Statistical Analysis 13: Comparison: V114 vs Prevenar 13™; GMC Ratio Serotype 23F: CI are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Other; GMC Ratio = 1.22, 95% CI 2-sided [1.07 to 1.40] — V114 / Prevenar 13™
Statistical Analysis 14: Comparison: V114 vs Prevenar 13™; GMC Ratio Serotype 22F: CI are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Other; GMC Ratio = 57.69, 95% CI 2-sided [51.20 to 65.00] — V114 / Prevenar 13™
Statistical Analysis 15: Comparison: V114 vs Prevenar 13™; GMC Ratio Serotype 33F: CI are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Other; GMC Ratio = 6.24, 95% CI 2-sided [5.46 to 7.14] — V114 / Prevenar 13™

9. Secondary Outcome: Percentage of Participants Who Meet Serotype-specific IgG Threshold Value of ≥0.35 μg/mL for Each Serotype at 30 Days PPS
Description: Sera from participants was used to measure vaccine-induced anti-PnPs serotype-specific IgG for the 15 serotypes using PnECL. The percentage of participants that achieve the threshold value of ≥0.35 μg/mL for each of the 13 serotypes shared by both V114 and Prevenar 13™ (Serotypes 1 to 23F); and the 2 serotypes unique to V114 (Serotypes 22F and 33F) was assessed.
Time Frame: 30 days PPS (Up to approximately study month 3)
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 588 | 591
Percentage of Participants
  Serotype 1: number analyzed (Participants) | 522 | 500
  Serotype 1 | 95.4 | 97.4
  Serotype 3: number analyzed (Participants) | 522 | 500
  Serotype 3 | 93.5 | 67.8
  Serotype 4: number analyzed (Participants) | 522 | 500
  Serotype 4 | 93.9 | 96.8
  Serotype 5: number analyzed (Participants) | 522 | 500
  Serotype 5 | 84.5 | 88.4
  Serotype 6A: number analyzed (Participants) | 522 | 500
  Serotype 6A | 73.2 | 92.6
  Serotype 6B: number analyzed (Participants) | 522 | 499
  Serotype 6B | 57.3 | 52.7
  Serotype 7F: number analyzed (Participants) | 522 | 500
  Serotype 7F | 97.9 | 99.0
  Serotype 9V: number analyzed (Participants) | 522 | 500
  Serotype 9V | 88.7 | 95.4
  Serotype 14: number analyzed (Participants) | 522 | 500
  Serotype 14 | 96.9 | 97.4
  Serotype 18C: number analyzed (Participants) | 522 | 500
  Serotype 18C | 92.3 | 93.0
  Serotype 19A: number analyzed (Participants) | 522 | 500
  Serotype 19A | 96.2 | 97.4
  Serotype 19F: number analyzed (Participants) | 522 | 500
  Serotype 19F | 98.9 | 99.4
  Serotype 23F: number analyzed (Participants) | 522 | 499
  Serotype 23F | 78.5 | 71.9
  Serotype 22F: number analyzed (Participants) | 522 | 500
  Serotype 22F | 95.6 | 5.2
  Serotype 33F: number analyzed (Participants) | 522 | 500
  Serotype 33F | 48.7 | 2.8
Statistical Analysis 1: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 1; Test type: Other; Percentage Difference = -2.0, 95% CI 2-sided [-4.4 to 0.3] — V114 minus Prevenar 13™; 95% CI are based on the Miettinen & Nurminen method
Statistical Analysis 2: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 3; Test type: Other; Percentage Difference = 25.7, 95% CI 2-sided [21.1 to 30.3] — V114 minus Prevenar 13™; 95% CI are based on the Miettinen & Nurminen method
Statistical Analysis 3: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 4; Test type: Other; Percentage Difference = -2.9, 95% CI 2-sided [-5.7 to -0.3] — V114 minus Prevenar 13™; 95% CI are based on the Miettinen & Nurminen method
Statistical Analysis 4: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 5; Test type: Other; Percentage Difference = -3.9, 95% CI 2-sided [-8.1 to 0.3] — V114 minus Prevenar 13™; 95% CI are based on the Miettinen & Nurminen method
Statistical Analysis 5: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 6A; Test type: Other; Percentage Difference = -19.4, 95% CI 2-sided [-23.9 to -15.0] — V114 minus Prevenar 13™; 95% CI are based on the Miettinen & Nurminen method
Statistical Analysis 6: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 6B; Test type: Other; Percentage Difference = 4.6, 95% CI 2-sided [-1.5 to 10.7] — V114 minus Prevenar 13™; 95% CI are based on the Miettinen & Nurminen method
Statistical Analysis 7: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 7F; Test type: Other; Percentage Difference = -1.1, 95% CI 2-sided [-2.9 to 0.5] — V114 minus Prevenar 13™; 95% CI are based on the Miettinen & Nurminen method
Statistical Analysis 8: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 9V; Test type: Other; Percentage Difference = -6.7, 95% CI 2-sided [-10.1 to -3.5] — V114 minus Prevenar 13™; 95% CI are based on the Miettinen & Nurminen method
Statistical Analysis 9: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 14; Test type: Other; Percentage Difference = -0.5, 95% CI 2-sided [-2.6 to 1.7] — V114 minus Prevenar 13™; 95% CI are based on the Miettinen & Nurminen method
Statistical Analysis 10: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 18C; Test type: Other; Percentage Difference = -0.7, 95% CI 2-sided [-3.9 to 2.6] — V114 minus Prevenar 13™; 95% CI are based on the Miettinen & Nurminen method
Statistical Analysis 11: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 19A; Test type: Other; Percentage Difference = -1.2, 95% CI 2-sided [-3.5 to 1.0] — V114 minus Prevenar 13™; 95% CI are based on the Miettinen & Nurminen method
Statistical Analysis 12: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 19F; Test type: Other; Percentage Difference = -0.5, 95% CI 2-sided [-2.0 to 0.7] — V114 minus Prevenar 13™; 95% CI are based on the Miettinen & Nurminen method
Statistical Analysis 13: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 23F; Test type: Other; Percentage Difference = 6.6, 95% CI 2-sided [1.3 to 11.9] — V114 minus Prevenar 13™; 95% CI are based on the Miettinen & Nurminen method
Statistical Analysis 14: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 22F; Test type: Other; Percentage Difference = 90.4, 95% CI 2-sided [87.4 to 92.7] — V114 minus Prevenar 13™; 95% CI are based on the Miettinen & Nurminen method
Statistical Analysis 15: Comparison: V114 vs Prevenar 13™; Percentage Difference: Serotype 33F; Test type: Other; Percentage Difference = 45.9, 95% CI 2-sided [41.3 to 50.3] — V114 minus Prevenar 13™; 95% CI are based on the Miettinen & Nurminen method

10. Secondary Outcome: Anti-PnPs Serotype-specific Opsonophagocytic Activity (OPA) GMTs for Each Serotype at 30 Days PTD
Description: Sera from participants was used to measure vaccine-induced anti-PnPs serotype-specific OPA using the multiplexed opsonophagocytic assay (MOPA). The GMT for each of the 13 serotypes shared by both V114 and Prevenar 13™ (Serotypes 1 to 23F); and the 2 serotypes unique to V114 (Serotypes 22F and 33F) was assessed. The within-group CIs were obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: 30 days PTD (Up to approximately study month 14)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 116 | 122
Titer
  Serotype 1: number analyzed (Participants) | 101 | 108
  Serotype 1 | 136.8 [107.2 to 174.6] | 164.6 [127.9 to 211.8]
  Serotype 3: number analyzed (Participants) | 98 | 103
  Serotype 3 | 321.5 [277.2 to 372.9] | 303.0 [253.2 to 362.6]
  Serotype 4: number analyzed (Participants) | 97 | 99
  Serotype 4 | 2231.7 [1770.5 to 2813.1] | 3206.4 [2626.6 to 3914.1]
  Serotype 5: number analyzed (Participants) | 102 | 108
  Serotype 5 | 791.6 [640.9 to 977.8] | 947.9 [784.3 to 1145.7]
  Serotype 6: number analyzed (Participants) | 98 | 99
  Serotype 6 | 3274.9 [2734.5 to 3921.9] | 5387.2 [4388.9 to 6612.5]
  Serotype 6B: number analyzed (Participants) | 94 | 95
  Serotype 6B | 2439.9 [1936.1 to 3074.7] | 3182.4 [2500.9 to 4049.7]
  Serotype 7F: number analyzed (Participants) | 97 | 100
  Serotype 7F | 6300.9 [5363.9 to 7401.7] | 10071.4 [8327.2 to 12181.0]
  Serotype 9V: number analyzed (Participants) | 97 | 103
  Serotype 9V | 1904.4 [1584.8 to 2288.4] | 2616.6 [2133.3 to 3209.4]
  Serotype 14: number analyzed (Participants) | 99 | 100
  Serotype 14 | 2633.8 [2102.6 to 3299.2] | 2582.1 [2089.5 to 3190.9]
  Serotype 18C: number analyzed (Participants) | 98 | 103
  Serotype 18C | 1968.6 [1676.4 to 2311.7] | 2091.8 [1789.1 to 2445.7]
  Serotype 19A: number analyzed (Participants) | 101 | 104
  Serotype 19A | 2995.6 [2556.5 to 3510.0] | 4254.3 [3649.3 to 4959.5]
  Serotype 19F: number analyzed (Participants) | 98 | 103
  Serotype 19F | 1793.9 [1535.3 to 2096.1] | 2012.3 [1677.0 to 2414.6]
  Serotype 23F: number analyzed (Participants) | 97 | 99
  Serotype 23F | 4517.8 [3685.1 to 5538.8] | 7987.6 [6149.3 to 10375.5]
  Serotype 22F: number analyzed (Participants) | 98 | 96
  Serotype 22F | 2405.2 [1980.5 to 2921.0] | 24.5 [16.0 to 37.7]
  Serotype 33F: number analyzed (Participants) | 96 | 101
  Serotype 33F | 14268.4 [11680.1 to 17430.2] | 1875.6 [1477.4 to 2381.3]

11. Secondary Outcome: Percentage of Participants Who Meet Serotype-specific OPA Threshold Value for Each Serotype at 30 Days PTD
Description: Sera from participants was used to measure vaccine-induced anti-PnPs serotype-specific OPA using the MOPA. The threshold dilution (% ≥) for each of the 13 serotypes shared by both V114 and Prevenar 13™ (Serotypes 1 to 23F) were as follows: 1:9, 1:19, 1:34, 1:27, 1:232, 1:40, 1:61, 1:151, 1:62, 1:115, 1:31, 1:113, 1:55. For Serotypes 22F and 33F the threshold dilution was 1:15 and 1:20 respectively. The within-group CIs were based on the exact binomial method of Clopper and Pearson.
Time Frame: 30 days PTD (Up to approximately study month 14)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 116 | 122
Percentage of Participants
  Serotype 1: number analyzed (Participants) | 101 | 108
  Serotype 1 | 95.0 [88.8 to 98.4] | 98.1 [93.5 to 99.8]
  Serotype 3: number analyzed (Participants) | 98 | 103
  Serotype 3 | 100.0 [96.3 to 100.0] | 98.1 [93.2 to 99.8]
  Serotype 4: number analyzed (Participants) | 97 | 99
  Serotype 4 | 100.0 [96.3 to 100.0] | 100.0 [96.3 to 100.0]
  Serotype 5: number analyzed (Participants) | 102 | 108
  Serotype 5 | 100.0 [96.4 to 100.0] | 100.0 [96.6 to 100.0]
  Serotype 6A: number analyzed (Participants) | 98 | 99
  Serotype 6A | 99.0 [94.4 to 100.0] | 100.0 [96.3 to 100.0]
  Serotype 6B: number analyzed (Participants) | 95 | 95
  Serotype 6B | 100.0 [96.2 to 100.0] | 100.0 [96.2 to 100.0]
  Serotype 7F: number analyzed (Participants) | 97 | 100
  Serotype 7F | 100.0 [96.3 to 100.0] | 100.0 [96.4 to 100.0]
  Serotype 9V: number analyzed (Participants) | 87 | 103
  Serotype 9V | 97.9 [92.7 to 99.7] | 100.0 [96.5 to 100.0]
  Serotype 14: number analyzed (Participants) | 99 | 100
  Serotype 14 | 100.0 [96.3 to 100.0] | 99.0 [94.6 to 100.0]
  Serotype 18C: number analyzed (Participants) | 98 | 103
  Serotype 18C | 100.0 [96.3 to 100.0] | 100.0 [96.5 to 100.0]
  Serotype 19A: number analyzed (Participants) | 101 | 104
  Serotype 19A | 100.0 [96.4 to 100.0] | 100.0 [96.5 to 100.0]
  Serotype 19F: number analyzed (Participants) | 98 | 103
  Serotype 19F | 100.0 [96.3 to 100.0] | 99.0 [94.7 to 100.0]
  Serotype 23F: number analyzed (Participants) | 97 | 99
  Serotype 23F | 100.0 [96.3 to 100.0] | 100.0 [96.3 to 100.0]
  Serotype 22F: number analyzed (Participants) | 98 | 96
  Serotype 22F | 99.0 [94.4 to 100.0] | 28.1 [19.4 to 38.2]
  Serotype 33F: number analyzed (Participants) | 96 | 101
  Serotype 33F | 100.0 [96.2 to 100.0] | 98.0 [93.0 to 99.8]

12. Secondary Outcome: Percentage of Participants Who Achieved the IgG Serotype-Specific Threshold Value of ≥0.35 μg/mL For Protocol Pre-Specified Serotypes at 30 Days PTD
Description: Sera from participants was used to measure vaccine-induced anti-PnPs serotype-specific IgG for the 15 serotypes using PnECL. As pre-specified in the protocol the percentage of participants from the two serotypes unique to V114 (Serotypes 22F and 33F) are presented, as well as the percentage of participants with the lowest response rate from any of the 13 shared serotypes randomized to Prevenar 13™ (Serotype 3).
Time Frame: 30 days PTD (Up to approximately study month 14)
Population: All randomized participants without deviations from the protocol that may substantially affect the results. For each pre-specified serotype, participants were only analyzed for the treatment group that they were randomized to.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 588 | 591
Percentage of Participants
  Serotype 22F: number analyzed (Participants) | 539 | 0
  Serotype 22F | 99.6 |
  Serotype 33F: number analyzed (Participants) | 539 | 0
  Serotype 33F | 99.1 |
  Serotype 3: number analyzed (Participants) | 0 | 537
  Serotype 3 |  | 83.8
Statistical Analysis 1: Comparison: V114 vs Prevenar 13™; Percentage Difference: V114 Serotype 22F minus Prevenar 13™ Serotype 3; Test type: Other — Percentage difference and CI are based on the Miettinen & Nurminen method; Percentage Difference = 15.8, 95% CI 2-sided [12.9 to 19.2] — V114 minus Prevenar 13™
Statistical Analysis 2: Comparison: V114 vs Prevenar 13™; Percentage Difference: V114 Serotype 33F minus Prevenar 13™ Serotype 3; Test type: Other — Percentage difference and CI are based on the Miettinen & Nurminen method; Percentage Difference = 15.3, 95% CI 2-sided [12.2 to 18.7] — V114 minus Prevenar 13™

ADVERSE EVENTS:
Time Frame: Non-serious AEs reported from Day 1 through 14 days following each vaccination. Serious AEs reported from Day 1 up to approximately study month 20. All-cause mortality (ACM) reported from randomization up to approximately study month 20.
Description: The ACM population was all randomized participants. For AEs the population was APaT, which consisted of participants who received at least 1 dose of study vaccination. The ACM and AEs for participants inadvertently vaccinated with both V114 and Prevenar 13™were reported separately from other participants.
Groups:
- V114 + Prevenar 13™: Participants inadvertently vaccinated with both V114 and Prevenar 13™
Arm/Group | V114 | Prevenar 13™ | V114 + Prevenar 13™
All-Cause Mortality (participants affected / at risk) | 0/591 | 0/593 | 0/1
Serious Adverse Events (participants affected / at risk) | 57/587 | 70/591 | 0/1
Other Adverse Events (participants affected / at risk) | 548/587 | 540/591 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=587) | Prevenar 13™ (N=591) | V114 + Prevenar 13™ (N=1)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 9 (11) | 10 (10) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Exanthema subitum (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Gastritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 8 (8) | 0 (0)
Gastroenteritis adenovirus (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis sapovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Otitis media acute (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Otitis media chronic (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 3 (3) | 3 (3) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 8 (8) | 5 (5) | 0 (0)
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Viral infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foreign body ingestion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Infantile spasms (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=587) | Prevenar 13™ (N=591) | V114 + Prevenar 13™ (N=1)
Diarrhoea (Gastrointestinal disorders) | 39 (48) | 45 (66) | 0 (0)
Injection site erythema (General disorders) | 266 (455) | 264 (443) | 1 (1)
Injection site induration (General disorders) | 246 (418) | 231 (392) | 0 (0)
Injection site pain (General disorders) | 238 (370) | 173 (257) | 0 (0)
Injection site swelling (General disorders) | 197 (315) | 174 (263) | 0 (0)
Pyrexia (General disorders) | 261 (447) | 251 (437) | 1 (1)
Rhinitis (Infections and infestations) | 29 (33) | 44 (51) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 8 (8) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 199 (354) | 198 (334) | 0 (0)
Somnolence (Nervous system disorders) | 271 (507) | 247 (473) | 0 (0)
Irritability (Psychiatric disorders) | 421 (1094) | 392 (1038) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/46/NCT04031846/Prot_SAP_000.pdf